CLINICAL TRIAL: NCT07386899
Title: Optimizing the Timing of Caffeinated Gum: Effects of 5- and 10-Minute Chewing on Plasma Caffeine Pharmacokinetics in Healthy Men
Brief Title: 5 vs 10-Minute Chewing of Caffeinated Gum: Plasma Caffeine Pharmacokinetics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Gülbin Rudarlı, Professor, Ege University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CAF-GUMPK-5v10-324S220
Record Dates: First submitted 2026-01-28; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Caffeine
Keywords: Pharmacokinetics; Plasma caffeine; Caffeinated chewing gum; Chewing duration; Absorption; Time to peak; Peak concentration; AUC
MeSH Terms: interventions — Caffeine

STUDY DESIGN:
Intervention Model Description: Two-condition, two-visit within-subject fixed-sequence crossover (5-min chewing at Visit 1; 10-min chewing at Visit 2), with ≥48 hours between visits.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 5-Minute Chewing (Experimental): Participants chew caffeinated chewing gum for 5 minutes (total caffeine approximately 300 mg).
  Interventions: Dietary Supplement: Caffeine 300 MG
- 10-Minute Chewing (Experimental): Participants chew caffeinated chewing gum for 10 minutes (total caffeine approximately 300 mg).
  Interventions: Dietary Supplement: Caffeine 300 MG

INTERVENTIONS:
Dietary Supplement: Caffeine 300 MG — 300 mg (three pieces; ~100 mg each) administered at each visit. Participants chew for 5 minutes in one condition and 10 minutes in the other condition.

SUMMARY:
The goal of this study is to understand how chewing duration affects how quickly caffeine from caffeinated chewing gum appears in the blood and how long higher caffeine levels are maintained. The study compares two chewing durations (5 minutes and 10 minutes) in healthy men.

Each participant attends two study visits on separate days at least 48 hours apart and completes both chewing conditions. At each visit, participants chew caffeinated gum that provides approximately 300 mg of caffeine. Blood samples are collected before chewing and at several time points for up to 3 hours after chewing to measure plasma caffeine levels.

Researchers will compare the two chewing durations to determine whether chewing time changes peak plasma caffeine concentration, the time to reach the peak, overall exposure over 0 to 180 minutes, and the time that plasma caffeine remains near the peak level. The results may help guide practical timing of caffeinated gum use.

DETAILED DESCRIPTION:
This is a within-subject, repeated-measures, two-visit, fixed-sequence study comparing two chewing durations of caffeinated gum (5 minutes vs 10 minutes). Participants attend two visits on separate days with at least 48 hours between visits to minimize carryover effects. The order is fixed: the 5-minute chewing condition is completed at Visit 1 and the 10-minute chewing condition at Visit 2.

At each visit, participants receive approximately 300 mg of caffeine via commercially available caffeinated chewing gum (three pieces; about 100 mg per piece). Venous blood samples are collected to measure plasma caffeine concentration over time. Samples are obtained at baseline (0 minutes), during chewing (5 minutes in both conditions and 10 minutes only in the 10-minute condition), and after chewing at 30, 50, 60, 80, 90, 120, and 180 minutes. Plasma caffeine is quantified using liquid chromatography-tandem mass spectrometry (LC-MS/MS).

The plasma caffeine concentration-time profile is used to derive pharmacokinetic outcomes, including peak plasma caffeine concentration, time to peak concentration, exposure from 0 to 180 minutes, and the duration that plasma caffeine remains at or above 90% and 80% of the individual peak concentration.

The study was approved by the Ege University Faculty of Medicine Medical Research Ethics Committee, and written informed consent was obtained from all participants prior to participation.

ELIGIBILITY:
Inclusion Criteria:

* Male, 18-35 years
* Good general health
* No regular use of medications or substances
* Habitual daily caffeine intake ≤300 mg/day

Exclusion Criteria:

* Habitual daily caffeine intake >300 mg/day
* Failure to participate in any study measurements
* Failure to comply with required test and measurement protocols
* Experiencing adverse effects from caffeine during the compliance period

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2025-04-22 (Actual); Primary Completion 2025-06-14 (Actual); Study Completion 2025-06-14 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Caffeine Concentration (Cpeak) | From baseline (0 minutes) up to 180 minutes post-chewing
  Highest observed plasma caffeine concentration over the 0-180 minute sampling period, quantified from venous blood samples analyzed by liquid chromatography-tandem mass spectrometry (LC-MS/MS). Unit: µg/mL.
Time to Peak Plasma Caffeine Concentration (Tpeak) | From baseline (0 minutes) up to 180 minutes post-chewing
  Time (minutes) from baseline (start of sampling) to the individual peak plasma caffeine concentration (Cpeak) within the 0-180 minute sampling period.
Area Under the Plasma Caffeine Concentration-Time Curve From 0 to 180 Minutes (AUC0-180) | 0 to 180 minutes post-chewing
  Total plasma caffeine exposure from 0 to 180 minutes calculated from measured plasma caffeine concentrations (trapezoidal method). Unit:mg·h/L.

SECONDARY OUTCOMES:
Duration Plasma Caffeine Remains at or Above 90% of Individual Peak (Sustain90) | 0 to 180 minutes post-chewing
  Duration (minutes) during which plasma caffeine concentration is at or above 90% of the individual Cpeak within the 0-180 minute sampling period.
Duration Plasma Caffeine Remains at or Above 80% of Individual Peak (Sustain80) | 0 to 180 minutes post-chewing
  Duration (minutes) during which plasma caffeine concentration is at or above 80% of the individual Cpeak within the 0-180 minute sampling period.
Plasma Caffeine Concentration-Time Profile | Baseline (0 minutes) through 180 minutes post-chewing
  Plasma caffeine concentrations (µg/mL) measured at prespecified time points: 0, 5, 10 (10-minute condition only), 30, 50, 60, 80, 90, 120, and 180 minutes post-chewing, analyzed by LC-MS/MS.

CONTACTS AND LOCATIONS:
Overall Officials: Hakan Arslan, Dr., Principal Investigator — Ege University; Gülbin Rudarlı, professor, Study Chair — Ege University
Locations (1):
- Ege University, Faculty of Sport Sciences, Izmir, Bornova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kamimori GH, Karyekar CS, Otterstetter R, Cox DS, Balkin TJ, Belenky GL, Eddington ND. The rate of absorption and relative bioavailability of caffeine administered in chewing gum versus capsules to normal healthy volunteers. Int J Pharm. 2002 Mar 2;234(1-2):159-67. doi: 10.1016/s0378-5173(01)00958-9. PMID 11839447